CLINICAL TRIAL: NCT06569771
Title: Evolution of the Patient's Perception of the Use of the Upper Limb After a Stroke During Intensive Rehabilitation
Acronym: ValetM-2024
Status: Recruiting | Type: Observational
Sponsor: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Other Study IDs: Perception Valet M 2024
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-08

CONDITIONS: Upper Limb Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering from motor impairment of the upper limbs following a stroke: Voluntary patients suffering from motor impairment of the upper limbs following a stroke
  Interventions: Diagnostic Test: Functional assessments

INTERVENTIONS:
Diagnostic Test: Functional assessments — * Computer Adaptive Test for Fugl-Meyer (CAT-FM)
  * Action Research Arm Test (ARAT)
  * Measurement of Functional Independence
  * Star cancellation test
  * Stroke Impact Scale
  * ACTIVLIM (assesses the ability to perform activities of daily living requiring the use of the upper limbs)

SUMMARY:
This study is being carried out in the context of rehabilitation after stroke, where persistent upper limb weakness is a major challenge. It aims to explore the relationship between observed function and patients' perceived participation in use.

ELIGIBILITY:
Inclusion Criteria:

* First stroke as defined by the World Health Organization.
* Upper limb paresis with a NIHSS National Institutes of Health Stroke Scale score > or = 1/4 for upper limb motor function

Exclusion Criteria:

* Life expectancy <12 months
* Inability to understand French.
* Pre-existing severe multiple disability affecting arm function.
* Presence of pre-existing central neurological pathologies.
* Mini-Mental State Examination < 21

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered a first stroke will be selected on transfer to a neurological rehabilitation service. They will be recruited on admission, provided they meet the inclusion and exclusion criteria.
  A combination of self-administered questionnaires and functional assessments will be carried out on the first day of multidisciplinary management in the neurological rehabilitation department and after two months in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess whether the perception of use of the impaired upper limb improves during intensive rehabilitation after a stroke. | Up to 2 months
  various tests : computer adaptive test F-M, ARA test, MIF test, star concellation test, ACTIVLIM test
To compare the difference between perception and observed function of the upper limb during intensive multidisciplinary rehabilitation treatment. | Up to 2 months
  various tests : computer adaptive test F-M, ARA test, MIF test, star concellation test, ACTIVLIM test

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Valet, MD, Principal Investigator — Grand Hôpital de Charleroi
Locations (2):
- Belgium (2):
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - CHU HELORA site Kennedy, Mons, Hainaut